CLINICAL TRIAL: NCT02195804
Title: A Phase I Open-label, Randomised, Single Dose, Three-way Crossover Relative Bioavailability Study of Ranitidine Hydrochloride (Maximum Strength ZANTAC 150®) Compared to Two Different 150 mg Ranitidine Hydrochloride Oral Disintegrating Tablet (ODT) Formulations Following Oral Administration in Fasting, Healthy Male Volunteers
Brief Title: Bioavailability Study of Ranitidine Hydrochloride (Maximum Strength ZANTAC 150®) Compared to Two Different 150 mg Ranitidine Hydrochloride Oral Disintegrating Tablet (ODT) in Fasting, Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1144.3
Record Dates: First submitted 2014-07-17; First posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Ranitidine

ARMS (3):
- Ranitidine HCL ODT Vanilla-Mint (Experimental)
  Interventions: Drug: Ranitidine hydrochloride ODT
- Ranitidine HCL ODT RM Vanilla-Mint (Experimental)
  Interventions: Drug: Ranitidine hydrochloride ODT RM
- Ranitidine HCL (Active Comparator): Maximum Strength ZANTAC 150®
  Interventions: Drug: Ranitidine hydrochloride

INTERVENTIONS:
Drug: Ranitidine hydrochloride ODT — Ranitidine hydrochloride ODT#1 150 mg (Vanilla-Mint)
  Arms: Ranitidine HCL ODT Vanilla-Mint
Drug: Ranitidine hydrochloride ODT RM — Ranitidine hydrochloride ODT Reduced Mannitol (RM) 150 mg Vanilla-Mint (ODT#2)
  Arms: Ranitidine HCL ODT RM Vanilla-Mint
Drug: Ranitidine hydrochloride
  Other Names: Maximum Strength ZANTAC 150®
  Arms: Ranitidine HCL

SUMMARY:
The objective of this study is to establish the relative bioavailability (BA) of two different ranitidine hydrochloride 150 mg ODT formulation in comparison to the current, over the counter (OTC) ranitidine hydrochloride (Maximum Strength ZANTAC 150®) formulation following oral single dose administration in fasting healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects based on: complete medical history, including a physical examination, vital signs (pulse rate (PR), systolic & diastolic blood pressure (BP) and body temperature), 12-lead electrocardiogram (ECG) and clinical laboratory tests
* Age ≥ 18 and Age ≤ 60 years
* BMI ≥ 18.5 and BMI ≤ 29.9 kg/m2 (Body Mass Index) and body weight of ≥ 55 kg
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

* Any clinically relevant abnormality found on the screening physical examination (including BP, PR) or ECG or in the opinion of the investigator the patient is not suitable for the study
* Any evidence of an acute or chronic gastrointestinal conditions or relevant concomitant medical disease
* History of acute porphyria
* History of peptic ulcer disease
* Heartburn requiring treatment (OTC or prescription medicine) within the last 30 days
* History of surgery of the gastrointestinal tract surgery (except appendectomy and cholecystectomy)
* History of relevant allergy / hypersensitivity (including allergy to H2 inhibitor) to the drug class, ranitidine hydrochloride or its excipients)
* Intake of prescription or over-the-counter (OTC) drugs with a long half-life (>24 hours) within at least 2 weeks or less than 10 half-lives of the respective drug prior to administration or during the trial
* Participation in another trial with an investigational drug within 30 days prior to administration or during the trial
* Inability to refrain from alcohol use 48 hours prior to drug administration until the end of the study visit for each treatment period
* History of alcohol (more than 60 g/day) or drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance as determined by the investigator
* Inability to comply with dietary regimen of trial site
* Subjects who test positive upon drug screening
* Subjects who consume caffeine or xanthine-containing drinks or foods (coffee, tea, cola, energy drinks, chocolate, etc.) 48 hours prior to study drug administration
* Subjects who consume citrus fruits and juices, (in particular grapefruits and Seville oranges, sour or bitter oranges), or products containing St. John's wort (Hypericum perforatum) are not allowed 7 days prior to dose administration
* Excessive physical activity or exercise (such as organized sports) during the trial period

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2009-05; Primary Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of ranitidine in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | up to 16 hours after drug administration
Maximum measured concentration of ranitidine in plasma (Cmax) | up to 16 hours after drug administration

SECONDARY OUTCOMES:
Area under the concentration-time curve of ranitidine in plasma over the time interval from 0 to the time of the last quantifiable data point (AUC0-tz) | up to 16 hours after drug administration
Time from dosing to the maximum concentration of ranitidine in plasma (tmax) | up to 16 hours after drug administration
Terminal rate constant in plasma (λz) | up to 16 hours after drug administration
Terminal half-life of ranitidine in plasma (t1/2) | up to 16 hours after drug administration
Mean residence time of the analyte in the body after po administration (MRTpo) | up to 16 hours after drug administration
Apparent clearance of the analyte in the plasma after extravascular administration (CL/F) | up to 16 hours after drug administration
Apparent volume of distribution during the terminal phase λz following an extravascular dose (Vz/F) | up to 16 hours after drug administration
Number of patients with adverse events | up to 38 days
Global assessment of tolerability by investigator on a 4-point scale | 24 hours after drug dosing at the end of each treatment period